CLINICAL TRIAL: NCT07164235
Title: Spondylodiscitis: a Retrospective Observational Study of the Alessandria University Hospital's Case Series.
Brief Title: Spondylodiscitis: a Retrospective Observational Study.
Acronym: SpAl
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: ASO.MInf.22.04
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Spondylodiscitis
Keywords: Spondylodiscitis; infectious processes; 18-FDG; 18 F-FDG-PET/CT
MeSH Terms: conditions — Discitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients diagnosed with spondylodiscitis — Patients admitted to the Infectious Diseases Department of the University Hospital of Alessandria between January 1, 2017, and December 31, 2024, who were diagnosed with spondylodiscitis

SUMMARY:
Spondylodiscitis is an infectious process affecting the vertebral bodies, intervertebral discs, and paraspinal tissues, sometimes involving the spinal cord, most often with a bacterial etiology. Instrumental diagnosis relies on CT, however, contrast-enhanced MRI is the most sensitive test for confirming the diagnosis, as abnormalities are usually detected earlier than with CT. More recently, nuclear diagnostics using 18-fluorodeoxyglucose (18-FDG) PET has proven very useful both for diagnosis and as a tool for monitoring therapeutic efficacy. Etiological diagnosis relies primarily on blood cultures and, if the former is not possible, diagnostic biopsy. Approximately one-third of patients lack a microbiological isolation, and the inability to implement targeted therapy is a known risk factor for treatment failure.

Therapeutic indications are giving way to shorter courses based on the use of oral medications, even though the epidemiology of the countries from which most of the clinical indications and literature originate is profoundly different from that of Italy. An epidemiological analysis of the cases referred to our Center is therefore of primary importance.

DETAILED DESCRIPTION:
Spondylodiscitis is an infectious process affecting the vertebral bodies, intervertebral discs, and paraspinal tissues, sometimes involving the spinal cord. The etiology is most often bacterial, with the main pathogens implicated being Staphylococcus aureus, streptococci, enterobacteriaceae, and other Gram-negative bacilli. Instrumental diagnosis relies on CT, which allows for the detection of lesions such as bony sequestrations and soft tissue abscesses, as well as the exclusion of epidural abscesses. Contrast-enhanced MRI, however, is the most sensitive test for confirming the diagnosis, as abnormalities are usually detected earlier than with CT.

More recently, nuclear imaging, particularly 18-fluorodeoxyglucose (18-FDG) PET, has proven very useful both for diagnosing tissue with high glucose metabolism and as a tool for monitoring therapeutic efficacy. 18F-FDG-PET/CT has been associated with greater accuracy than MRI in diagnosing early spondylodiscitis in the first 2 weeks after symptom onset. Another important advantage of 18F-FDG-PET/CT over MRI is the potential identification of metastatic infectious foci, especially in patients with bacteremia, allowing for rapid source control. 18F-FDG-PET/CT is also useful for spondylodiscitis caused by mycobacteria, fungi, or Brucella, with some data suggesting different uptake values depending on the etiology.

Etiological diagnosis, however, relies primarily on blood cultures, which can be positive in up to 50% of cases of native spondylodiscitis caused by S. aureus. When noninvasive isolation is not possible, a diagnostic biopsy is necessary. Despite the use of invasive techniques, approximately one-third of patients lack microbiological isolation, and the inability to implement targeted therapy is a known risk factor for treatment failure. It also leads to the use of broad-spectrum antimicrobials, with environmental and sometimes economic consequences.

Therapeutic indications, until now based on case series and cohort studies dating back more than 40 years, are giving way to shorter courses based on the use of orally administered drugs. However, the epidemiology of the countries from which most of the clinical indications and literature on bone infections originate is profoundly different from that of Italy. Therefore, an epidemiological analysis of the cases referred to our Center is of primary importance.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female subjects aged ≥ 18 years;
* Diagnosis of spondylodiscitis confirmed radiologically and microbiologically
* Admission to Infectious Diseases Unit between January 1, 2017 and December 31, 2024
* Signed informed consent.

Exclusion Criteria:

* Age <18 years
* Lack of signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient will be taken from adult male or female population aged ≥ 18 years, who received diagnosis of spondylodiscitis confirmed radiologically and microbiologically and who was admitted to Infectious Diseases Unit between January 1, 2017 and December 31, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Descriptive analysis | Baseline
  Description of the characteristics of patients diagnosed with spondylodiscitis admitted to the University Hospital of Alessandria from 2017 to 2024

SECONDARY OUTCOMES:
Pre- and post-pandemic comparison of clinical and management characteristics of patients with spondylodiscitis | Baseline
  Comparison of the differences in the characteristics of patients hospitalized before and after 06/03/2020 (pre-pandemic and post-pandemic period)
Comparison of the differences between patients with confirmed and unconfirmed microbiological diagnosis | Baseline
  Evaluate any differences in duration between patients with a confirmed and unconfirmed microbiological diagnosis of spondylodiscitis
Concordance between PET results and antibiotic therapy | Baseline
  Evaluate the concordance between PET results and antibiotic therapy discontinuation in the absence of relapse at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center SC Infrastruttura Ricerca Formazione Innovazione Dipartimento Attività Integrate Ricerca e Innovazione Azienda Ospedaliero-Universitaria SS Antonio e Biagio e C. Arrigo di Alessandria, Alessandria, Piedmont, Italy